CLINICAL TRIAL: NCT06505642
Title: Combined Needle-based Confocal Laser Endomicroscopy Cone-Beam Computed Tomography Navigation Bronchoscopy: a Proof of Principle Study
Brief Title: NCLE-Cone-beam CT Navigation Bronchoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. J.T. Annema, MD, PhD, Prof. dr. Jouke Annema, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86502.018.24
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-08

CONDITIONS: Lung Neoplasm; Peripheral Lung Parenchyma Tumor; Lung Cancer
Keywords: Confocal Laser Endomicroscopy; Bronchoscopy; Cone beam computed tomography; Image guided bronchoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nCLE + CBCT-NB (Experimental): Patients with a suspected malignant peripheral pulmonary nodule(s) referred for cone beam ct navigation bronchoscopy for tissue sampling.
  Interventions: Device: needle-based confocal laser endomicroscopy

INTERVENTIONS:
Device: needle-based confocal laser endomicroscopy — needle-based confocal laser endomicroscopy at the tip of the TBNA needle for two punctures, combined with confirmatory CBCT spin for tool-in-lesion confirmation
  Other Names: cone beam computed tomography navigation bronchoscopy

SUMMARY:
The goal of this proof of principle observational study is to investigate in patients with suspected peripheral pulmonary nodules. The main question it aims to answer is:

• What is the concordance between CBCT navigation success (tool-in-lesion on CBCT spin) and nCLE tool-in-lesion confirmation (tool-in-lesion nCLE criteria observed).

Participants scheduled to undergo a diagnostic conebeam navigation bronchoscopy will be included in the study. nCLE imaging at the tip of the TBNA needle will be added to the procedure for study purposes.

Two needle punctures of the pulmonary nodule will be followed by nCLE imaging directly followed by a tool-in-lesion CBCT spin in order to compare nCLE results with CBCT results.

DETAILED DESCRIPTION:
Lung cancer remains a significant problem in current society with one of the higher cancer related mortality rates. The increased use of chest computed tomography (CT) and the po-tential future lung cancer screening result in an increased detection of early-stage peripheral lung cancer. Bronchoscopies are often indicated to collect tissue for diagnosis and to aid treatment decision making.

Diagnostic bronchoscopy for peripheral lung nodules remains challenging despite many tech-nological innovations. The procedure comprises three essential pillars needed for a diagnos-tic success: navigation to the lesion, tool-in-lesion confirmation and adequate tissue retrieval.

Cone beam computed tomography navigation bronchoscopy (CBCT-NB) is a fairly new tech-nique that provides coarse navigation to the pulmonary lesion with real-time guidance using augmented fluoroscopy (AF). An initial CBCT scan allows for segmentation of the target le-sion and selecting the optimal pathway. Repeated CBCT scanning allows for confirmation that the target has been reached (navigation success) or if repositioning is needed.

Although the technique is very promising, an often discussed disadvantage of CBCT is the inherent use of ionizing radiation, limited availability and challenges with small nodules lo-cated in the basal and posterior fields due to respiratory motion. Most procedures ask for multiple CBCT spins both for trajectory planning, tool adjustments and tool-in-lesion confir-mation. This, combined with extensive use of fluoroscopy is associated with radiation expo-sure for both patients and the investigation team. Additionally, CBCT-NB with AF provides information from a global perspective rather than a local perspective. In experienced centers, coarse navigation guidance seems of lesser concern and fine positioning and optimal tissue sampling are the biggest problems to be overcome. The persistently low diagnostic yield of navigation bronchoscopies can for the majority be attributed mispositioning of the tools in "the last centimeter". Therefore there is a need for complementary techniques providing real-time information for fine-tuning the needle position such as needle-based confocal laser en-domicroscopy (nCLE) also called the "smart needle".

Confocal laser endomicroscopy (CLE) is a high-resolution microscopic technique that visual-izes individual cells in real-time at the tip of the biopsy needle, allowing for real-time micro-scopic feedback for fine tuning needle positioning and tool-in-lesion confirmation. Currently, it is unknown which (combination of) techniques are the most optimal (i.e., leading to a high di-agnostic yield and cost-effective). Therefore, research is needed to investigate the potential of new (combinations of) techniques. To date, there are no reports on the combination of CBCT-NB with nCLE.

Objective: This study aims to investigate proof of principle of utilizing nCLE during CBCT-NB navigation bronchoscopy. A confirmatory CBCT spin is considered the gold standard for tool-in-lesion but is associated with additional radiation exposure. The aim is to investigate the concordance between CBCT navigation success (tool-in-lesion on CBCT spin) and nCLE tool-in-lesion confirmation (tool-in-lesion nCLE criteria observed). The investigators also hypothesize that nCLE could reduce or replace the need for additional confirmatory CBCT scans and limit fluoroscopy use.

Study design: Investigator-initiated proof of principle medical device study

Study population: Patients (18 years and older) with (suspected) pulmonary nodules with an indication for cone-beam computed tomography navigation bronchoscopy.

Procedure: Cone beam computed tomography navigation bronchoscopy combined with needle-based confocal laser endomicroscopy.

Main study parameters/endpoints:

* CBCT-NB navigation success as either tool-in-lesion OR unsuccessful
* nCLE tool-in-lesion confirmation, defined as tool-in-lesion nCLE criteria observed

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Suspected pulmonary nodule with an indication for CBCT-NB (decided by multidisciplinary tumour board)
* Nodule must be solid or partially solid
* Solid part of the nodule must be at least 8 mm
* Largest dimension of the nodule on CT equal or less than 30 mm
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Inability or non-willingness to provide informed consent
* Patients with an endobronchial visible lung tumor on bronchoscopic inspection
* Patients in which the target lesion is within reach of the linear EBUS scope
* Lung nodules that resolved at the time of index intraprocedural CBCT
* Failure to comply with the study protocol
* Patients with known allergy for fluorescein or risk factors for an allergic reaction
* Pregnant or breastfeeding women
* Patients with hemodynamic instability
* Patients with refractory hypoxemia
* Patients with a therapeutic anticoagulant that cannot be held for an appropriate in-terval before the procedure
* Patients who are unable to tolerate general anesthesia according to the anesthesiologist
* Patient undergoing chemotherapy as several chemotherapies have fluorescent properties at the same wavelength (e.g. doxorubicin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
CBCT navigation success and nCLE tool-in-lesion confirmation | Intra-procedure
  CBCT-NB navigation success: tool-in-lesion OR unsuccessful navigation nCLE tool-in-lesion confirmation: in-lesion nCLE criteria seen

SECONDARY OUTCOMES:
Technical feasibility | Intra-procedure
  Proportion of nCLE imaging that are successful (meaning that the preloaded needle can be advanced through the working channel, puncture the nodule, advance the CLE probe and start imaging) resulting good quality images.
Safety | Up to 7 days post procedure
  Number and proportion of (severe) adverse events ((S)AEs) and investigational procedure related adverse events (AEs)
Diagnostic yield | up to 6 months post procedure
  Proportion (expressed in percentages) of patients in whom the bronchoscopic procedure results in a definitive diagnosis out of the total number of patients that have received the diagnostic bronchoscopic procedure.
Diagnostic sensitivity for malignancy | up to 6 months post procedure
  Proportion (expressed in percentages) of patients that have malignancy diagnosed by bronchoscopic tissue sampling, relative to the total number of patients with a final diagnosis of malignancy as determined by the reference standard.
Sensitivity, specificity and accuracy of real-time nCLE imaging assessment | Intra-procedure
  Sensitivity, specificity and accuracy of real-time nCLE imaging assessment all described in percentages.
Sensitivity, specificity and accuracy of post-procedure nCLE image assessment | Intra-procedure
  Sensitivity, specificity and accuracy of post-procedure nCLE image assessment described as percentages.
Interobserver agreement (IOA) and intraobserver reliability (IOR) | Intra-procedure
  Interobserver agreement (IOA) represented by the Cohen's kappa statistics (mean with 95% confidence intervall) and intraobserver reliability (IOR) represented by the Cohen's kappa statistics (mean +/- standard deviation)

OTHER OUTCOMES:
Total procedure duration | Intra-procedure
  Total procedure duration in minutes (introduction brochoscope to removal of bronchoscope)

CONTACTS AND LOCATIONS:
Overall Officials: Jouke Annema, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided